CLINICAL TRIAL: NCT03764215
Title: An Open Label, Phase Ib Study to Evaluate the Impact of Low Doses of Nilotinib Treatment on Safety, Tolerability and Biomarkers in Huntington's Disease
Brief Title: Nilotinib in Huntington's Disease
Acronym: Tasigna HD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Karen E. Anderson, MD, Director, Huntington Disease Care, Education and Research Center at MedStar Georgetown University Hospital and Georgetown University Medical Center, Georgetown University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0440
Record Dates: First submitted 2018-11-27; First posted 2018-12-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — nilotinib

STUDY DESIGN:
Intervention Model Description: Ten (10) participants will receive an oral dose of 150mg Nilotinib once daily for 3 months (group 1). If this dose is tolerated another 10 participants will receive an oral dose of 300mg Nilotinib once daily (group 2) for 3 months.
Masking Description: We propose to perform an open label, Phase Ib, proof of concept study to evaluate the impact of low doses of Nilotinib treatment on safety, tolerability and biomarkers in participants with HD. We propose an adaptive design based on safety and tolerability of 150mg Nilotinib treatment for 3 months. We will first enroll 10 participants who will receive an oral dose of 150mg Nilotinib once daily (group 1) for 3 months. If these participants tolerate 150mg dose of Nilotinib, an additional 10 new HD participants (group 2) will be enrolled to evaluate the effects of 300 mg dose of Nilotinib for 3 months. We will then compare baseline with the effects of 3-months Nilotinib treatment within each group and between groups (1 and 2). Participants (group 1 and 2) will return for a follow up visit one month after the termination of 3-months treatment with Nilotinib and results will compared to baseline visits and end of study visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Ten (10) participants will receive an oral dose of 150mg Nilotinib once daily for 3 months (group 1). If Nilotinib 150 mg per mouth daily dose is tolerated by the 1st group of 10 participants for 3 months, another 10 participants will receive an oral dose of 300mg Nilotinib once daily (group 2) for 3 months.
  Interventions: Drug: Nilotinib 150 MG

INTERVENTIONS:
Drug: Nilotinib 150 MG — 10 participants will receive an oral dose of 150mg Nilotinib once daily for 3 months (group 1). If this dose is tolerated another 10 participants will receive an oral dose of 300mg Nilotinib once daily (group 2) for 3 months.

SUMMARY:
Based on strong pre-clinical evidence of the effects of Nilotinib on neurodegenerative pathologies, including autophagic clearance of neurotoxic proteins, neurotransmitters (dopamine and glutamate), immunity and behavior, the investigators conducted an open label pilot clinical trial in mid-to-advanced PD with dementia (PDD) and Dementia with Lewy Bodies (DLB) (stage 3-4) patients. Participants (N=12) were randomized 1:1 to once daily oral dose of 150mg and 300mg Nilotinib for 6 months. The investigators data suggests that Nilotinib penetrates the brain and inhibits CSF Abelson (Abl) activity via reduction of phosphorylated Abl in agreement with pre-clinical data. Several studies suggest that CSF alpha-Synuclein and Abeta42 are decreased and CSF total Tau and p-Tau are increased in PD and DLB. The investigators data shows attenuation of loss of CSF alpha-Synuclein and Abeta40/42 with 300mg (50% of the CML dose) compared to 150mg Nilotinib after 6 months treatment. CSF homovanillic acid (HVA), which is a by-product of dopamine metabolism, is significantly increased; and CSF total Tau and p-Tau are significantly reduced (N=5, P<0.05) with 300mg Nilotinib between baseline and 6 months treatment. Despite the reduction of L-Dopa replacement therapies in our study, the Unified Parkinson's Disease Rating Scale (UDPRS) I-IV scores improved with 150mg (3.5 points) and 300mg (11 points) from baseline to 6 months and worsened (13.7 points and 11.4 points) after 3 months withdrawal of 150mg and 300mg, respectively. Other non-motor functions e.g. constipation was resolved in all patients and cognition was also improved (3.5 points) using both the Mini-Mental Status Exam (MMSE) or the Scales for Outcomes in Parkinson's Disease-Cognition (SCOPA-Cog) between baseline and 6 months. MMSE scores returned to baseline after 3 months of Nilotinib withdrawal. These data are very compelling to evaluate the effects of Nilotinib in an open label proof-of-concept study in patients with HD.

DETAILED DESCRIPTION:
The investigators performed an open label phase I clinical trial using two commercially available doses of Nilotinib (150 and 300mg capsules) in patients with advanced PDD and DLB. These indications have some overlapping pathologies and clinical symptoms and share common plasma and CSF biomarkers, including alpha-Synuclein, Abeta42/40, total Tau and p-Tau. The investigators obtained preliminary data showing that Nilotinib crosses the BBB and is detected in the CSF, suggesting Abl inhibition and downstream target engagement (alpha-Synuclein, Tau and Abeta) in the CNS (pharmacodynamics). Nilotinib increased CSF HVA levels as a downstream biomarker of dopamine metabolism. These data provide feasibility to test Nilotinib in a phase Ib clinical trial to demonstrate safety, tolerability and changes in disease biomarkers in patients with HD. The Huntingtin gene provides the genetic information for a protein that is also called "huntingtin" (Htt). Expansion of CAG (cytosineadenine-guanine) triplet repeats in the gene coding for the Huntingtin protein results in an abnormal protein, mutant Htt (mHTT), which gradually leads to protein accumulation within neurons and neuronal cell damage. Based on preclinical and clinical studies, the investigators hypothesize that Nilotinib will be safe and tolerable in individuals with HD. The level of HVA is significantly reduced in HD patients compared to controls (22), and the investigators expect Nilotinib to increase HVA levels. Nilotinib may also affect CSF level of total Huntingtin proteins and cell death markers, including NSE and S100B. The investigators further hypothesize that the investigators may see evidence of change in cognitive, motor or behavioral outcomes that will help us to build a better clinical development program going forward.

Neurodegenerative diseases, including HD, are a group of genetic and sporadic disorders associated with neuronal death and progressive nervous system dysfunction. Cancer is also a collection of related genetic diseases, in which cells begin to divide without stopping and spread into surrounding tissues. Unlike neurodegeneration, in which no regeneration happens when damaged or aging postmitotic neurons die, damaged cells survive when they should die in cancer, resulting in uncontrolled mitotic cell division to form tumors. Cancerous tumors are malignant as they spread or invade nearby tissues by cellular contiguity or metastasize via blood and/or humoral transport. In neurodegeneration, the spread of disease by contiguity is supported by the hypotheses that toxic or "prion-like" proteins propagate along neuroanatomical pathways leading to progressive spread of disease and cell death. In neurodegeneration, failure of cellular quality control mechanisms leads to inadequate protein degradation via the proteasome or autophagy, resulting in intracellular accumulation of neurotoxic proteins. Consequently, these proteins are secreted from a pre-synaptic neuron and can traverse the synaptic cleft and enter a contiguous post-synaptic neuron. Secreted proteins may not penetrate an adjacent cell via the synapse but they may be re-routed into the cell and recycled via the endosomal system to fuse with autophagic vacuoles like the autophagosome or the lysosome. Microglia, the brain resident immune cells may also phagocytose and destroy toxic proteins. Accumulation of neurotoxic proteins, including alpha-Synuclein (Lewy bodies), beta-amyloid plaques, Tau tangles, Huntingtin, prions and TDP-43 are major culprits in neurodegeneration. These toxic proteins trigger progressive apoptotic cell death leading to loss of many central nervous system (CNS) functions, including mentation, cognition, language, movement, gastrointestinal motility, sleep and many others. The discoveries of toxic protein propagation from cell to cell, leading to progression of neurodegeneration triggered a series of pre-clinical and clinical studies to limit protein propagation via antibodies (active and passive immune therapies) that can capture the protein and destroy it en route to healthy neurons. This approach is fraught with difficulties, including failure to arrest neurocognitive decline and brain edema/inflammation. Manipulation of autophagy is a novel therapeutic approach that focuses on degradation of neurotoxic proteins at the manufacturing site in order to prevent their secretion and propagation. This novel strategy leads to unclogging the cell's disposal machine and degradation of toxic proteins, thus preserving neuronal survival via bulk digestion of abnormal proteins. Preservation of neuronal survival maintains the level of neurotransmitters that are necessary for cognitive, motor and other CNS functions, leading to alleviation of symptoms as well as arrest of neurodegeneration. As neurons are post-mitotic cells, pulsatile autophagy may promote protein degradation and provide an effective disease-modifying therapy for neurodegenerative diseases. Autophagy is a double-edged sword in cancer, either preventing accumulation of damaged proteins and organelles to suppress tumors, or promoting cell survival mechanisms that lead to tumor growth and proliferation. Leukemia and many other cancer treatments have been revolutionized by manipulation of autophagy, which leads to bulk degradation of unwanted or toxic molecules. For example in leukemia, genetic mutations and DNA damage can lead to large numbers of abnormal white blood cells (leukemia cells and leukemic blast cells) to accumulate in the blood and bone marrow, crowding out normal blood cells. Autophagy can lead to the degradation of the products of cancer-causing genes (oncogenes), tumor suppressor genes, damaged DNA and essential components of the cytosol, thereby controlling abnormal mitotic division and limiting tumor growth. Autophagy can also lead to self-cannibalization via promotion of programmed cell death, or apoptosis. Activation of the tumor suppressor p53 in response to DNA damage leads the cell to arrest proliferation, initiate DNA repair, and promote survival. However, if the DNA damage cannot be resolved by p53, it can trigger apoptotic death. Cell division and apoptosis are mediated by signaling mechanisms via the endosomal (early and recycling) system. Tyrosine kinases are activated via auto phosphorylation, triggering various signaling mechanisms that mediate cell division and/or apoptosis. Tyrosine kinase inhibition via de-phosphorylation leads to signaling via the late endosomal-lysosomal pathway, thus increasing autophagic degradation and tumor growth. TKIs have significantly improved the life quality and expectancies in many cancers, including CML. CML is characterized by the translocation of chromosomes 9 and 22 to form the "Philadelphia" chromosome resulting in the expression of a constitutively active Breakpoint Cluster Region-Abelson (BCR-Abl) tyrosine kinase. This oncogenic protein activates intracellular signaling pathways and induces cell proliferation. Our laboratory investigated TKIs that activate autophagy and are FDA-approved for CML, thus significantly reducing research and development efforts and cost by re-purposing for new indications. Abl is activated in neurodegeneration. A fraction of Nilotinib crosses the blood-brain-barrier (BBB), inhibits Abl and facilitates autophagic amyloid clearance, leading to neuroprotection and improved cognition and motor behavior. Mice treated with a much lower dose of these drugs (<25% of the typical CML dose) show significant motor and cognitive improvement and degradation of alpha-Synuclein, beta-amyloid, Tau and TDP-43 without evidence of increased inflammation. There was also significant reversal of neurotransmitter alterations, including dopamine and glutamate in several models of neurodegeneration. As a modulator of myeloid cells, Nilotinib may also positively regulate neuronal death and produce neuro-restorative effects via increased production of necessary growth factors and proliferation of myeloid-derived glia. Autophagic toxic protein clearance and production of growth factors may restore loss of neurotransmitters, leading to improved motor and cognitive functions. Nilotinib provides a double-edge sword via manipulation of autophagy to inhibit cell division and tumor growth in CML on one hand, and promote toxic protein degradation and neuronal survival in neurodegeneration on the other hand. The investigators propose to perform an open label, Phase Ib, proof of concept study to evaluate the impact of low doses of Nilotinib treatment on safety, tolerability and biomarkers in participants with HD. The investigators propose an adaptive design based on safety and tolerability of 150mg Nilotinib treatment for 3 months. The investigators will first enroll 10 participants who will receive an oral dose of 150mg Nilotinib once daily (group 1) for 3 months. If these participants tolerate 150mg dose of Nilotinib, i.e. with no exacerbation of chorea and behavioral symptoms and no other AEs (i.e. myelosuppression, QTc prolongation, liver/pancreatic toxicity, etc ), an additional 10 new HD participants (group 2) will be enrolled to evaluate the effects of 300 mg dose of Nilotinib for 3 months. The investigators will then compare baseline with the effects of 3-months Nilotinib treatment within each group and between groups (1 and 2). Participants (group 1 and 2) will return for a follow up visit one month after the termination of 3-months treatment with Nilotinib and results will compared to baseline visits and end of study visits. Ten (10) participants will receive an oral dose of 150mg Nilotinib once daily for 3 months (group 1). If this dose is tolerated another 10 participants will receive an oral dose of 300mg Nilotinib once daily (group 2) for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Capable of providing informed consent and complying with study procedures. Subjects who are unable to provide consent may use a Legally Authorized Representative (LAR).
* Patients between the age of 25-90 years, medically stable
* Clinical diagnosis of HD with either a confirmed family history or positive CAG repeat (CAG≥35)
* MoCA ≥ 22
* Able to perform the TMT-B in ≤240 seconds
* Total Functional Capacity 7-12
* Stable concomitant medical and/or psychiatric illnesses, in the judgement of the PI.
* QTc interval 350-460 ms, inclusive
* Participants must be willing to undergo LP at baseline and 3 months after treatment

Exclusion Criteria:

* Patients with hypokalemia, hypomagnesaemia, or long QT syndrome- QTc≥461 ms
* Concomitant drugs known to prolong the QTc interval and history of any cardiovascular disease, including myocardial infarction or cardiac failure, angina, arrhythmia
* History or presence of cardiac conditions including:

  1. Cardiovascular or cerebrovascular event (e.g. myocardial infarction, unstable angina, or stroke)
  2. Congestive heart failure
  3. First, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances
  4. Any history of Torsade de Pointes
* Treatment with any of the following drugs at the time of screening or the preceding 30 days, and/or planned use over the course of the trial:

  1. Treatment with Class IA or III antiarrhythmic drugs (e.g. quinidine)
  2. Treatment with QT prolonging drugs (www.crediblemeds.org)- excluding Selective Serotonin Reuptake Inhibitors (SSRIs) (e.g. Citalopram, Escitalopram, Paroxetine, Sertraline, Duloxetine, Trazodone, etc.)
  3. Strong CYP3A4 inhibitors (including grapefruit juice). The concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) must be avoided. Grapefruit products may also increase serum concentrations of Nilotinib. Should treatment with any of these agents be required, therapy with Nilotinib should be interrupted.
  4. Anticoagulants, including Coumadin (warfarin), heparin, enoxaparin, daltiparin, xarelto, etc.
  5. St. John's Wort and the concomitant use of strong other CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital) must be avoided since these agents may reduce the concentration of Nilotinib.
* Abnormal liver function defined as AST and/or ALT > 100% the upper limit of the normal
* Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal
* History of HIV, clinically significant chronic hepatitis, or other active infection
* Females must not be lactating, pregnant or with possible pregnancy
* Medical history of liver or pancreatic disease
* Clinical signs indicating syndromes other than idiopathic PD, including corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, Babinski sign

  .Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any active major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality
* Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history of skin melanoma or stable prostate cancer are not exclusionary)
* Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder
* Must not be on any immunosuppressant medications (e.g. IVig)
* Must not be enrolled as an active participant in another clinical study

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing any Adverse events and Serious Adverse Events | 3 months
  will be measured using the occurrence of adverse events (AEs) and serious adverse events (SAEs) deemed to be possibly, probably, or definitely related to the study drug. AEs of interest are defined as QTc prolongation, myelosuppression, hepatotoxicity and pancreatitis as listed in Table 1. These AEs will be tracked over the course of the trial and reviewed by the data and safety monitoring board (DSMB) at scheduled meetings and in real time. SAEs and AEs are known to be related to drug use at 800mg daily in cancer. A small safety trial using lower oral daily doses of 150 mg and 300 mg Nilotinib in 12 PD patients showed one cardiac SAE over a six-month treatment period. Based on preliminary clinical data, investigator's brochure (IB) and scheduled EKGs and lab tests, SAEs and AEs will be evaluated real-time and on case-by-case basis.
CSF levels of biomarkers linked to Disease symptoms Chorea and behavioral symptoms | 3 months
  Prior studies from our group showed that Nilotinib treatment increases the CSF levels of HVA, suggesting alteration of dopamine level. We will evaluate the effects of potential changes of dopamine levels on Chorea and behavioral symptoms in HD participants. We will use an adaptive study design that will allow examination of the effects of 150mg Nilotinib once daily in 10 HD participants. If participants in this group do not exhibit worsening chorea or behavioral changes, then 300mg Niloitnib will be given to a new group of 10 additional participants. These potential AEs will be tracked over the course of the trial and reviewed by the DSMB at scheduled meetings and in real time.
Number of participants tolerating the drug by the ability of remaining on treatment | 3 months
  for a given participant will be defined as the ability of participants to remain on treatment. Overall tolerability of the drug will be defined as an acceptable number of up to 25% discontinuations.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Pagan F, Hebron M, Valadez EH, Torres-Yaghi Y, Huang X, Mills RR, Wilmarth BM, Howard H, Dunn C, Carlson A, Lawler A, Rogers SL, Falconer RA, Ahn J, Li Z, Moussa C. Nilotinib Effects in Parkinson's disease and Dementia with Lewy bodies. J Parkinsons Dis. 2016 Jul 11;6(3):503-17. doi: 10.3233/JPD-160867. PMID 27434297
- See also: Translational Neurotherapeutics Program at Georgetown University Medical Center — https://neurology.georgetown.edu/translational_neurotherapeutics